CLINICAL TRIAL: NCT05234346
Title: An Open-Label, Pilot Study to Evaluate the Safety, Tolerability, and Efficacy of 5-ALA-Phosphate + SFC as an Immune System Enhancer Along With Vaccination Against SARS-CoV-2 Virus Infection
Brief Title: ALACOVID Study for Vaccinated Subjects
Acronym: COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PH/210904/5ALP/COVID
Record Dates: First submitted 2022-02-05; First posted 2022-02-10 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-05

CONDITIONS: COVID-19 Respiratory Infection
MeSH Terms: interventions — Sodium Glutamate

STUDY DESIGN:
Intervention Model Description: An Open-Label, Pilot Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 150 mg 5-ALAPhosphate + SFC (Experimental): 2 capsules in the morning after breakfast (before 11 AM) and 1 capsule in the evening after a snack or after dinner (before 8 PM) orally with water for 21 days.
  Interventions: Drug: 150 mg 5-ALAPhosphate + SFC
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 150 mg 5-ALAPhosphate + SFC — 2 capsules in the morning after breakfast (before 11 AM) and 1 capsule in the evening after a snack or after dinner (before 8 PM) orally with water for 21 days.
  Arms: 150 mg 5-ALAPhosphate + SFC
Other: Placebo — No Description for the intervention
  Arms: Placebo

SUMMARY:
In this study, it is hypothesized that administration of 5-ALA-Phosphate + SFC in subjects vaccinated against Covid-19 could contribute in enhancing the targeted function of the immune system, which might lead to re-activation and/or increase of the vaccination response. Thus, in the present study, we will be evaluating the safety and efficacy of 5-ALA-Phosphate + SFC in subjects receiving the Covid-19 vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Male & female aged ≥ 18 years and ≤70 years.
2. Subjects with documented proof of 1st dose of vaccination within 3 months of planned 2nd dose. (If government of India implements booster dose then subjects needs to have a documented proof of 2nd dose)
3. Subjects planning to have 2nd /3rd dose of COVID-19 vaccine (Covishield/ Covaxin). (If government of India implements booster dose then subjects planning to have a 3rd dose of vaccine will be included in this study)
4. Subject willing and able to provide a written informed consent

Exclusion Criteria:

1. Subjects with anemia (male: <12 g/dl, females: <11 g/dl)
2. Subjects with more than 2.5 times upper limit of ALT & AST parameters.
3. Subjects not willing to stop intake of any vitamin/s or mineral/s supplements during the trial except for those allowed in the study.
4. Subjects with acute symptomatic COVID-19 infection indicated by fever, dry cough and severe respiratory distress.
5. Subjects with SpO2 < 90%.
6. Subjects with history of genetic disorders.
7. Subjects with history of:

   1. Anaphylactic or allergic reaction to a previous dose of COVID-19 vaccine
   2. Immediate or delayed-onset anaphylaxis or allergic reaction to vaccines or injectable therapies, pharmaceutical products, food-items etc.
8. Pregnancy & Lactation:

   a. Pregnant & Lactating women have not been part of any COVID-19 vaccine clinical trial so far. Therefore, women who are pregnant or not sure of their pregnancy; and lactating women should not receive COVID-19 vaccine at this time
9. Provisional / temporary contraindications:

   1. Persons having active symptoms of SARS-CoV-2 infection.
   2. SARS-COV-2 patients who have been given anti-SARS-CoV-2 monoclonal antibodies or convalescent plasma
   3. Signs of acute infection or illness
   4. Hospitalized patients due to any illness.
10. Subjects with known history (diagnosed case) of porphyria, or chronic serious liver disease, kidney disease or heart problems.
11. Subjects with frequent complaints of cold, fever, cough.
12. Subjects with irritable bowel syndrome.
13. Subjects who are frequent travelers or are planning to travel.
14. Subject has demonstrated previous intolerance of 5-ALA and/or SFC by topical or oral administration.
15. Subjects with known allergy to 5-ALA containing foods (spinach, shitake mushroom, octopus, baker's yeast, wine, vinegar, sake less).
16. Subjects on vitamin D supplements
17. Males and females of reproductive potential who have not agreed to use an adequate method of contraception during the study

    1. For females, adequate birth control methods will be defined as: hormonal contraceptives, intrauterine device or double barrier contraception, i.e., condom

       + diaphragm, condom or diaphragm + spermicidal gel or foam.
    2. For males, adequate birth control methods will be defined as double barrier contraception, i.e., condom + diaphragm, condom or diaphragm + spermicidal gel or foam.
    3. For females, menopause is defined as one year without menses; if in question, a follicle-stimulating hormone of >40 U/ml must be documented. Hysterectomy, bilateral oophorectomy, or bilateral tubal ligation must be documented, as applicable.
18. Subjects who are unable or unwilling to comply with requirements of the clinical trial.
19. Participation in any other clinical trial of an experimental treatment for COVID-19.
20. Subjects having any other family member participating in this study.
21. Subjects who may be excluded at the Investigator's discretion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-06-18 (Actual); Study Completion 2022-06-18 (Actual)

PRIMARY OUTCOMES:
Adverse product reaction | Day 0
  To determine the safety of 21 days oral administration of 5-ALA-Phosphate + SFC in subjects vaccinated with COVID-19 vaccine.
Adverse product reaction | Day 1
  To determine the safety of 21 days oral administration of 5-ALA-Phosphate + SFC in subjects vaccinated with COVID-19 vaccine.
Adverse product reaction | Day 7
  To determine the safety of 21 days oral administration of 5-ALA-Phosphate + SFC in subjects vaccinated with COVID-19 vaccine.
Adverse product reaction | Day 21
  To determine the safety of 21 days oral administration of 5-ALA-Phosphate + SFC in subjects vaccinated with COVID-19 vaccine.

SECONDARY OUTCOMES:
Absolute change in GMT of IgG levels against Covid-19 spike protein | Day 0 and Day 21
  Elecsys Anti-SARS-CoV-2 S kit will be used to measure the levels of IgG post vaccination on baseline and at the end of the study (day 21).
European Quality of Life Five Dimension Five level questionnaire | Day 0 , Day 1, Day 7 and Day 21
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The subject is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the subject's health state. The Lower level is denoted as 1 and the highest level is denoted as 5. The EQ-5D-5L QoL questionnaire will be completed by the subject.
World Health Organization Well-Being Index questionnaire | Day 0 , Day 1, Day 7 and Day 21
  The 5-item World Health Organization Well-Being Index (WHO-5) is a short and generic global rating scale measuring subjective well-being.
Visual Analogue Scale for pain and fatigue | Day 0 , Day 1, Day 7 and Day 21
  The subjects is asked to place a line perpendicular to the VAS line at the point that represents their current situation for pain and fatigue (question 4). Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity

CONTACTS AND LOCATIONS:
Locations (4):
- India (4):
  - BAJ RR Hospital and Research Centre, Dombivali, Maharashtra
  - Leelawati Care Hospital-Nasik (SMO), Nashik, Maharashtra
  - Ranka Hospital, Pune, Maharashtra
  - JNU Institute for Medical Sciences and Research Centre, Jaipur, Rajasthan